CLINICAL TRIAL: NCT05945628
Title: Human Hippocampal Contributions to Rapid Encoding-retrieval Interactions During Memory Formation
Brief Title: Basic Experimental Study of Hippocampal Memory Functions
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IRB22-1300; 1R01MH128552 (NIH)
Record Dates: First submitted 2023-06-27; First posted 2023-07-14 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Memory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Experiment 1 (Experimental): Subjects with iEEG electrodes implanted will perform an eye-tracking memory task in which they view pictures of naturalistic scenes and later undergo memory testing for these scene pictures. For the memory test, studied scenes will be repeated and presented along with novel (foil) scenes. Subjects will attempt to discriminate studied from novel scenes using button press responses. Eye movements will be remotely (noninvasively) tracked using a camera during both study and test. This memory task will take about 1.5 hours to complete. 20 subjects undergoing iEEG recordings as part of epilepsy treatment will be assigned to this study experiment condition.
  Interventions: Behavioral: Different cognitive and memory demands during the memory experiment
- Experiment 2 (Experimental): Subjects with iEEG electrodes implanted will perform an eye-tracking memory task in which they view arrays of everyday objects arranged as a grid and later undergo memory testing for these object image arrays. Half of the object-image arrays are studied actively (subjects view objects in any order they wish) and half are studied passively (viewing patterns are predetermined and subjects must follow along). For the memory test, subjects attempt to pick studied objects from among novel (foil) objects and replace them at studied locations using the computer mouse. Eye movements will be remotely (noninvasively) tracked using a camera during the study phases. This memory task will take about 1.5 hours to complete. 20 subjects undergoing iEEG recordings as part of epilepsy treatment will be assigned to this study experiment condition.
  Interventions: Behavioral: Different cognitive and memory demands during the memory experiment
- Experiment 3 (Experimental): The same 20 subjects with iEEG electrodes implanted who perform Study Experiment Condition 2 will perform the same eye-tracking memory task described for Study Experiment Condition 1. For these subjects, high-frequency electrical stimulation will be delivered through the iEEG electrodes on a subset of study trials, with half of stimulated trials receiving stimulation of the hippocampus and the other half receiving stimulation of the amygdala. This memory task will take about 1.5 hours to complete and will be performed on a different day of their inpatient visit than the procedures for Study Experiment Condition 2.
  Interventions: Behavioral: Different cognitive and memory demands during the memory experiment; Other: Different electrical stimulation parameters during cognitive and memory demands
- Experiment 4 (Experimental): The same 20 subjects with iEEG electrodes implanted who perform Study Experiment Condition 1 will perform the same eye-tracking memory task described for Study Experiment Condition 2. For these subjects, high-frequency electrical stimulation will be delivered through the iEEG electrodes on a subset of study trials, with half of stimulated trials receiving stimulation of the hippocampus and the other half receiving stimulation of the amygdala. This memory task will take about 1.5 hours to complete and will be performed on a different day of their inpatient visit than the procedures for Study Experiment Condition 1.
  Interventions: Behavioral: Different cognitive and memory demands during the memory experiment; Other: Different electrical stimulation parameters during cognitive and memory demands
- Experiment 5 (Experimental): Subjects with iEEG electrodes implanted will perform the same eye-tracking memory task as described for Study Experiment Condition 1. This is a different group of iEEG subjects selected based on having iEEG electrodes implanted in the hippocampus as well as in at least one location of the Dorsal Attention Network (DAN), which is a region of interest for the experiment condition. 20 subjects undergoing iEEG recordings as part of epilepsy treatment will be assigned to this study experiment condition.
  Interventions: Behavioral: Different cognitive and memory demands during the memory experiment
- Experiment 6 (Experimental): The same group of 20 iEEG subjects that are included in Study Experiment Condition 5 will perform the same eye-tracking memory task as described for Study Experiment Condition 2. This experiment condition will be performed on a different day of the inpatient visit than participation in Study Experiment Condition 5.
  Interventions: Behavioral: Different cognitive and memory demands during the memory experiment

INTERVENTIONS:
Behavioral: Different cognitive and memory demands during the memory experiment — Study conditions will involve attempting to memorize visual scenes, attempting to memorize arrays of visual objects, viewing in a self-directed manner, viewing in a passive other-directed manner, and making memory judgments about whether stimuli are studied versus novel.
Other: Different electrical stimulation parameters during cognitive and memory demands — Study conditions will involve different parameters for electrical stimulation delivered through iEEG electrodes, including the presence of stimulation (no stimulation versus stimulation) and the location of stimulation (hippocampus versus amygdala).
  Arms: Experiment 3; Experiment 4

SUMMARY:
This project tests the role of the human hippocampus in providing online representation of episodic content and providing the top-down signals to brain networks for visuospatial attention and visual processing needed to drive visual sampling for the formation of coherent episodic memories. This hypothesis will be tested in several experiments that measure and manipulate hippocampal activity within eye-tracking tasks designed to isolate the interplay between memory and visual sampling during memory formation. These experiments will be performed in individuals with epilepsy undergoing neurosurgical procedures as part of clinical care, as this provides invasive recordings of neural activity (intracranial electroencephalography, or "iEEG") from the hippocampus and other regions of interest with temporal resolution that matches the rapid pace of eye movements. The temporal resolution of iEEG is key to addressing the hypotheses concerning how the hippocampus drives visual sampling, in addition to responding to it. Direct electrical stimulation through the iEEG electrodes will also be used to test the necessary role of hippocampal processing in driving active visual sampling. By rigorously testing the role of hippocampus in interaction with large-scale networks during the process of memory formation that occurs via active sampling, this project aims to better understand mechanisms relevant to the disruptions of memory formation that occur in neurological and psychiatric disorders.

DETAILED DESCRIPTION:
This is a basic experimental study performed with human subjects (BESH) that seeks to understand the mechanisms by which the human hippocampus supports visual sampling during episodic memory formation. Research subjects will be assigned to one of six study experiment conditions that each uses different experimental procedures to test a different portion of the mechanistic hypotheses that are the focus of the study. All of the study conditions involve memory experiments performed during eye-movement tracking, with different methods used to assess brain activity during standardized laboratory conditions in relation to the experimental task. Subjects will perform the experiments while their brain activity is recorded via intracranial EEG (iEEG), which is being performed for clinical purposes as part of epilepsy treatment unrelated to the experimental objectives.

Study Experiment Condition 1: Subjects with iEEG electrodes implanted will perform an eye-tracking memory task in which they view pictures of naturalistic scenes and later undergo memory testing for these scene pictures. For the memory test, studied scenes will be repeated and presented along with novel (foil) scenes. Subjects will attempt to discriminate studied from novel scenes using button press responses. Eye movements will be remotely (noninvasively) tracked using a camera during both study and test. This memory task will take about 1.5 hours to complete. 20 subjects undergoing iEEG recordings as part of epilepsy treatment will be assigned to this study experiment condition.

Study Experiment Condition 2: Subjects with iEEG electrodes implanted will perform an eye-tracking memory task in which they view arrays of everyday objects arranged as a grid and later undergo memory testing for these object image arrays. Half of the object-image arrays are studied actively (subjects view objects in any order they wish) and half are studied passively (viewing patterns are predetermined and subjects must follow along). For the memory test, subjects attempt to pick studied objects from among novel (foil) objects and replace them at studied locations using the computer mouse. Eye movements will be remotely (noninvasively) tracked using a camera during the study phases. This memory task will take about 1.5 hours to complete. 20 subjects undergoing iEEG recordings as part of epilepsy treatment will be assigned to this study experiment condition.

Study Experiment Condition 3: The same 20 subjects with iEEG electrodes implanted who perform Study Experiment Condition 2 will perform the same eye-tracking memory task described for Study Experiment Condition 1. For these subjects, high-frequency electrical stimulation will be delivered through the iEEG electrodes on a subset of study trials, with half of stimulated trials receiving stimulation of the hippocampus and the other half receiving stimulation of the amygdala. This memory task will take about 1.5 hours to complete and will be performed on a different day of their inpatient visit than the procedures for Study Experiment Condition 2.

Study Experiment Condition 4: The same 20 subjects with iEEG electrodes implanted who perform Study Experiment Condition 1 will perform the same eye-tracking memory task described for Study Experiment Condition 2. For these subjects, high-frequency electrical stimulation will be delivered through the iEEG electrodes on a subset of study trials, with half of stimulated trials receiving stimulation of the hippocampus and the other half receiving stimulation of the amygdala. This memory task will take about 1.5 hours to complete and will be performed on a different day of their inpatient visit than the procedures for Study Experiment Condition 1.

Study Experiment Condition 5: Subjects with iEEG electrodes implanted will perform the same eye-tracking memory task as described for Study Experiment Condition 1. This is a different group of iEEG subjects selected based on having iEEG electrodes implanted in the hippocampus as well as in at least one location of the Dorsal Attention Network (DAN), which is a region of interest for the experiment condition. 20 subjects undergoing iEEG recordings as part of epilepsy treatment will be assigned to this study experiment condition.

Study Experiment Condition 6: The same group of 20 iEEG subjects that are included in Study Experiment Condition 5 will perform the same eye-tracking memory task as described for Study Experiment Condition 2. This experiment condition will be performed on a different day of the inpatient visit than participation in Study Experiment Condition 5.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+ years old
* Native English speakers.
* Normal or corrected-to-normal near and far vision.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-01-16 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
iEEG theta band power | Outcome assessed 5 minutes after intervention
  iEEG is used to measure slow and fast theta power
iEEG phase synchrony to eye movement | Outcome assessed 5 minutes after intervention
  iEEG is used to measure phase synchronization of theta to eye movements

SECONDARY OUTCOMES:
Eye movements | Outcome assessed 5 minutes after intervention
  Eye movements are recorded during task performance using a remote camera and analyzed based on the location of gaze and the pattern of gaze among screen location regions of interest
Memory task performance | Outcome assessed 5 minutes after intervention
  Subjects attempt to discriminate studied from novel (foil) scenes and object images and to recall the spatial locations of objects. Outcome measure is recall performance

CONTACTS AND LOCATIONS:
Overall Officials: Joel Voss, PhD, Principal Investigator — University of Chicago
Locations (2):
- United States (2):
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared through the National Institute of Mental Health (NIMH) Data Archive
Supporting Information: SAP, Analytic Code
Time Frame: Data will become available starting July 2023
Access Criteria: Individuals with an NIMH Data Archive account may request access to the de-identified data